CLINICAL TRIAL: NCT07017309
Title: Feasibility and Preliminary Efficacy of a Telerehabilitation Protocol for Diastasis Recti Abdominis: A Pilot Study
Brief Title: Telerehabilitation for Diastasis Recti
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Anastasia Skoura, PhD candidate, University of Patras
Other Study IDs: DRATelerehab-Pilot-16331
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diastasis Recti; Telerehabilitation; Diastasis Recti Abdominis (DRA); Diastasis Recti And Weakness Of The Linea Alba
Keywords: Diastasis recti abdominis; postpartum rehabilitation; telerehabilitation; core stabilization; Pelvic Floor Exercises; Women's Health Physiotherapy
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group
  Interventions: Behavioral: Telerehabilitation Protocol for Diastasis Recti

INTERVENTIONS:
Behavioral: Telerehabilitation Protocol for Diastasis Recti — 12-week telerehabilitation program combining synchronous (live, supervised by physiotherapists) and asynchronous (video -recorded) therapeutic exercise sessions focused on progressive inner core exercises (i.e. transversus abdominis, pelvic floor muscle retraining), outer core strengthening, and functional retraining.

SUMMARY:
This is a pilot study exploring how a 12-week telerehabilitation program can help new mothers manage diastasis recti abdominis (DRA)-a common trunk dysfunction which causes abdominal muscle separation after childbirth. Instead of needing to attend in-person sessions, participants are encouraged to join guided exercise sessions online, with real-time supervision from a physiotherapist. The study aims to assess participant satisfaction with the remote program using a standardized questionnaire. It also evaluates potential changes in abdominal muscle separation (diastasis) through ultrasound, improvements in trunk muscle endurance using functional tests, and changes in body image perception using a body image questionnaire.

DETAILED DESCRIPTION:
This pilot study investigates the feasibility, patient satisfaction, and preliminary clinical effects of a 12-week telerehabilitation program targeting postpartum women diagnosed with diastasis recti abdominis (DRA). The intervention is delivered remotely and combines synchronous (real-time, supervised by physiotherapists) and asynchronous (video-recorded) therapeutic exercise sessions. Participants are required to attend two synchronous sessions per week via teleconference, which allows for real-time supervision and interaction with a specialized physiotherapist. They are also encouraged to attend one additional session per week independently using pre-recorded content. The exercise protocol includes progressive-load training focusing on inner core activation (i.e. transversus abdominis, pelvic floor muscles), outer core strengthening, and functional retraining.

Assessments are conducted at baseline, week 4, week 8, and post-intervention (week 12). Ultrasound imaging is used to measure inter-recti distance (IRD) at standard anatomical locations (2 cm above, 5 cm above, and 2 cm below the umbilicus) at baseline and post-intervention. Trunk muscle endurance is assessed through established functional tests, including curl-up manoeuvre, plank variations and McGill's trunk flexor endurance test at baseline, week 4, week 8, and post-intervention (week 12). Body image is evaluated using a validated Greek version of the Body Image States Scale (BISS_Greek) both at baseline and at the end of the intervention. Patient satisfaction is measured via the Greek version of the Telehealth Usability Questionnaire (TUQ_Greek), also accompanied by a custom-designed satisfaction question. Adherence is tracked using exercise diaries.

The study complies with ethical standards in accordance with the Declaration of Helsinki and has been approved by the Research Ethics Committee (R.E.C.) of the University of Patras (Internal Code: 16331/29-01-2024). All participants receive comprehensive written information about the study and data protection procedures and provide informed consent prior to participation. Patient data are anonymized and stored securely on a coded cloud-based platform accessible only to authorized research team members. Any adverse events are managed appropriately, documented in detail, and medical consultation is available during assessment and rehabilitation hours.

Missing, inconsistent, or uninterpretable data are addressed through imputation methods. A comprehensive data dictionary has been developed to ensure consistency in variable definitions, coding, and expected ranges. The accuracy and completeness of data entries is ensured by the research team through internal data validation and comparison with source data.

Participants are recruited through multiple channels, including posters and leaflets distributed at the University of Patras, the University General Hospital of Patras, and throughout the wider Achaia region. Recruitment is also supported by professional networks such as the Panhellenic Medical Association, the Panhellenic Physiotherapists' Association, and individual healthcare professionals (e.g., gynecologists, urologists, obstetricians, surgeons), public engagement events are organized across the Achaia region, and study information are promoted via the university website (Department of Physiotherapy), social media, and professional conferences.

Given the exploratory nature of this pilot study, no formal power calculation has been conducted. The sample size is intended to assess feasibility and inform the design of future larger-scale trials. Descriptive statistics will summarise participant characteristics and satisfaction outcomes. Repeated-measures ANOVA or non-parametric equivalents will be used to analyze changes over time in clinical outcomes, depending on data distribution. Statistical significance is set at p<0.05

ELIGIBILITY:
Inclusion Criteria:

* female volunteers aged 18 - 50
* with established DRA (IRD ≥ 2.8 cm) according to Mota et al., (2018) criteria
* at least 6 months postpartum
* able to voluntarily contract the transversus abdominis and pelvic floor muscles - comfortable with digital technology and having access to a smartphone, tablet, or computer with a camera and internet connection

Exclusion Criteria:

* recent abdominal surgery (excluding cesarean section)
* having given birth less than 6 months prior to participation
* serious musculoskeletal disorders limiting exercise participation
* neurological conditions limiting exercise participation
* chronic respiratory disease limiting exercise participation
* connective tissue disorders that could affect the structure of the linea alba
* body mass index (BMI) ≥ 30 kg/m²

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Participants from the wider Achaia region in Greece are invited to join the study through informational leaflets and posters placed in key locations such as the University Campus and the University General Hospital of Patras, as well as through social media channels. Additionally, details about the study are shared by local professional associations and healthcare providers-including obstetricians, midwives, and surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Telehealth Usability Questionnaire | Assessed at 12 weeks (end of intervention)
  Telehealth Usability Questionnaire is a validated tool including 21 items that assess six domains: usefulness, ease of use and learnability, interface quality, interaction quality, reliability, satisfaction and future use. Items are rated on a 7-point Likert scale, from "1: strongly disagree" to "7: strongly agree", and with higher average scores indicating greater usability. Maximum score can be 7, while minimum score can be 1.
Satisfaction Assessment | Assessed at 12 weeks (end of intervention)
  A closed-ended question, asking participants to rate their satisfaction with the telerehabilitation program on a 5-point Likert scale, from 1 : "not at all satisfied" to 5 "very satisfied."Higher values on the scale indicate higher satisfaction.

SECONDARY OUTCOMES:
Inter-recti distance (IRD) | Measured at baseline, and at 12 weeks (end of intervention)
  IRD is assessed using a real-time 2D diagnostic ultrasound imaging unit at three locations; at 2 cm and 5 cm above the umbilicus and at 2 cm below the umbilicus, in a supine, relaxed position with knees flexed and during exhalation.
Trunk flexion endurance | Measured at baseline, week 4, week 8, and at 12 weeks
  Trunk flexion endurance is assessed in a static trunk flexion position on a mat, using a stopwatch and is documented in seconds. Higher values indicate higher endurance.
Front plank endurance | Measured at baseline, week 4, week 8, and at 12 weeks
  Front plank endurance is assessed in a front plank position on a mat, using a stopwatch and is documented in seconds. Higher values indicate higher endurance.
Right side plank endurance | Measured at baseline, week 4, week 8, and at 12 weeks
  Right side plank endurance is assessed in a right side plank position on a mat, using a stopwatch and is documented in seconds. Higher values indicate higher endurance.
Left side plank endurance | Measured at baseline, week 4, week 8, and at 12 weeks
  Left side plank endurance is assessed in a left side plank position on a mat, using a stopwatch and is documented in seconds. Higher values indicate higher endurance.
McGill's Trunk Flexor Endurance Test | Measured at baseline, week 4, week 8, and at 12 weeks
  McGill's Trunk Flexor Endurance Test is assessed in an inclined sitting position on a mat, using a stopwatch and is documented in seconds. Higher values indicate higher endurance.
Body Image Assessment (BISS) | Measured at baseline, and at 12 weeks (end of intervention)
  The questionnaire consists of six statements related to how individuals perceive their physical appearance, body size and shape, weight, feelings of physical attractiveness, as well as current feelings about appearance compared to usual perceptions. Responses are rated on a 9-point bipolar Likert scale. A higher total score indicates a higher body image perception.
Adherence | Assessed at 12 weeks (end of intervention)
  Participant adherence is tracked by recording the number and type (remote supervised, or video-based) of weekly exercise sessions using a custom-made exercise diary. Higher numbers indicate higher adherence. Highest total number of sessions is 36 (up to 24 can be supervised sessions and up to 12 can be video recorded sessions). At least 24 sessions (both supervised and video-recorded) are required for inclusion in the final analysis. Minimum total number of sessions is 24.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, PhD, Study Director — University of Patras
Locations (1):
- Laboratory of Clinical Rehabilitation and Research (CPRlab), University of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No